CLINICAL TRIAL: NCT01133470
Title: An Open Label, Balanced, Randomized, Two-way, Single Dose, Crossover Bioequivalence Study of Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tabs of Dr. Reddy's and Allegra-D 24 hr ER Tabs of Aventis, in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tablets of Dr. Reddy's and Allegra D 24 Hour ER Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. Indu Bhushan / Senior Director, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-VIN-029
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Fexofenadine Hydrochloride + Pseudoephedrine Hydrochloride
MeSH Terms: interventions — fexofenadine; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fexofenadine HCl + Pseudoephedrine HCl (Experimental): Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tablets of Dr. Reddy's Laboratories
  Interventions: Drug: Fexofenadine HCl + Pseudoephedrine HCl
- Allegra-D 24 hour ER Tablets (Active Comparator): Allegra-D 24 hour ER Tablets of Aventis Pharmaceuticals INC., USA.
  Interventions: Drug: Fexofenadine HCl + Pseudoephedrine HCl

INTERVENTIONS:
Drug: Fexofenadine HCl + Pseudoephedrine HCl — Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tablets of Dr. Reddy's KLaboratories Limited
  Other Names: Allegra-D 24 hour ER Tablets

SUMMARY:
The purpose of this study is to

1. Compare and evaluate the single dose, crossover, bioequivalence study of Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tablets and Allegra-D 24 hr tablets.
2. Monitor the adverse events and ensure the safety of subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover bioequivalence study of Fexofenadine HCl 180 mg + Pseudoephedrine HCl 240 mg ER Tablets of Dr. Reddy's and Allegra-D 24 hour ER Tablets of Aventis Pharmaceuticals Inc., USA in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Human subjects aged between 18 and 45 years (including both)
* Subjects'weight within the normal range according to normal values for the Body Mass Index (18.5 to 24.9kgm2)with minimum of 50 kg weight.
* Subjects with normal health as determined by personal medical history clinical examination and laboratory examinations within the clinically acceptable normal range.
* Subjects having normal 12-lead electrocardiogram (ECG).
* Subjects having normal chest X-Ray (P/A view).
* Have a negative urine screen for drugs of abuse (including amphetamines,barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Have negative alcohol breath test.
* Subjects willing to adhere to the protocol requirements and to provide written informed consent.

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any of the following criteria:

* Hypersensitivity to Fexofenadine Hydrochloride and Pseudoephedrine Hydrochloride or related drugs.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 10 cigarettes or beedi's/day).
* History or presence of significant asthma, urticaria or other allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumour.
* History or presence of cancer.
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg.
* Diastolic blood pressure less than SO mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°F or more than 98.5°F.
* Respiratory rate less than 12/minute or more than 20/minute
* SUbjects who have used any prescription medication, within 14 days of period 01 dosing or OTC medication within 14 days of period 01 dosing.
* Major illness during 3 months before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Subjects who have consumed xanthine-containing products (including caffeine, theobromines, etc.) within 48 hours prior to period 01 dosing.
* Subjects who have consumed food or beverages containing grapefruit or pomelo within 14 days prior to period 01 dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2007-02; Primary Completion 2007-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dharmesh Domadia, Principal Investigator — Veeda Clinical Research Pvt. Ltd.,
Locations (1):
- Veeda Clinical Research Pvt. Ltd.,, Ahmedabad, Gujarat, India